CLINICAL TRIAL: NCT05442177
Title: Clinical Observation of Integrated Chinese Medicine With Western Medicine for the Reduction of Chemotherapy-induced Hematologic Toxicity
Status: Completed | Type: Observational
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Chia-Ying Chuang, Chinese medicine department, Taichung Tzu Chi Hospital
Other Study IDs: REC104-12
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Myelosuppression
Keywords: Traditional Chinese Medicine; radial pulse assessment; sphygmography; pulse diagnosis; myelosuppression; cancer
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Chemotherapy and Integrated Chinese Medicine With Western Medicine for cancer treatment

SUMMARY:
We conducted an observational study to investigate the effectiveness and safety of Integrated Chinese Medicine With Western Medicine for bone marrow suppression induced by chemotherapy in patients with cancer. The TCM constitution and pulse diagnosis was also observed in the study.

DETAILED DESCRIPTION:
Patients with cancer under chemotherapy and integrated Western and Chinese medicine were enrolled in this observational study. The assessment of radial pressure pulse (RPP) was performed before and after chemotherapy. The correlation between the spectral energy (SE0-10 Hz, SE10-50 Hz, and SE13-50 Hz) of the RPP at six diagnosis positions and the blood cell counts before and after chemotherapy were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer diagnosed through pathological histology
* Patients with cancer under chemotherapy and Integrated Chinese Medicine With Western Medicine
* Patients with an Eastern Cooperative Oncology Group Performance score of 0-2
* Patients having normal liver and kidney functions and electrocardiography and eligible for chemotherapy with normal bone marrow hematopoietic function
* Patients who were voluntarily involved in this study

Exclusion Criteria:

* Cases that did not meet the inclusion criteria
* Patients who could not cooperate with pulse diagnosis
* Patients with underlying diseases such as chronic obstructive pulmonary disease, cardiac failure, chronic renal failure, cirrhosis, etc.
* Patients with severe infection
* Patients with severe cachexia

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cancer under chemotherapy and Integrated Chinese Medicine With Western Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Chemotherapy-induced Hematologic Toxicity | one month
  the blood cell count before and after chemotherapy was collected for measurement of severity of myelosuppression